CLINICAL TRIAL: NCT05691465
Title: A Phase II Study of Lutetium Lu 177 Dotatate in Metastatic Prostate Cancer With Neuroendocrine Differentiation
Brief Title: Testing the Safety and Effectiveness of Radiation-based Treatment (Lutetium Lu 177 Dotatate) for Metastatic Prostate Cancer That Has Neuroendocrine Cells
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-05173; NCI-2022-05173 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10487 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10487 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2023-01-18; First posted 2023-01-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Prostate Adenocarcinoma With Neuroendocrine Differentiation; Metastatic Prostate Neuroendocrine Carcinoma; Metastatic Prostate Small Cell Neuroendocrine Carcinoma; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Ga(III)-DOTATOC; gallium Ga 68 dotatate; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lutetium Lu 177 dotatate) (Experimental): Patients receive lutetium Lu 177 dotatate IV over 30 minutes. Cycles repeat Q6W for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive gallium Ga 68-dotatate IV during screening then undergo PET/CT scan at baseline and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Gallium Ga 68-DOTATATE; Drug: Lutetium Lu 177 Dotatate; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Gallium Ga 68-DOTATATE — Given IV
  Other Names: (68)Ga-DOTA-TATE; 68Ga-DOTA-0-Tyr3-Octreotate; 68Ga-DOTATATE; Gallium Ga 68 Oxodotreotide; Gallium Oxodotreotide Ga-68; Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium (177Lu) Oxodotreotide; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial studies how well lutetium Lu 177 dotatate works in treating patients with prostate cancer with neuroendocrine differentiation that has spread to other places in the body (metastatic). Neuroendocrine differentiation refers to cells that have traits of both hormone-producing endocrine cells and nerve cells. These cells release hormones into the blood in response to a signal from the nervous system. Hormones are biological substances that circulate through the bloodstream to control the activity of other organs or cells in the body. Lutetium Lu 177-dotatate is a radioactive drug. It binds to a protein called somatostatin receptor, which is found on some neuroendocrine tumor cells. Lutetium Lu 177-dotatate builds up in these cells and gives off radiation that may kill them. It is a type of radioconjugate and a type of somatostatin analog. Treatment with Lutetium Lu 177 dotatate may shrink the tumor in a way that can be measured in patients with metastatic prostate cancer with neuroendocrine differentiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the objective response rate at 6 months for patients treated with lutetium Lu 177 dotatate using Prostate Cancer Working Group (PCWG) 3 criteria.

SECONDARY OBJECTIVES:

I. Evaluate the 6-month radiographic progression-free survival of neuroendocrine-differentiated prostate cancer treated with lutetium Lu 177 dotatate.

II. Determine if the change in fludeoxyglucose (FDG)-positron emission tomography (PET) signal from pre-treatment to after 2 doses of lutetium Lu 177 dotatate correlates with objective response rate.

EXPLORATORY OBJECTIVES:

I. Evaluate the potential to perform patient-specific dosimetry of lutetium Lu 177 dotatate using gamma imaging to predict treatment response and renal toxicity.

II. Perform gene expression analysis of circulating tumor cells to identify pre-treatment biomarkers of response and signatures of resistance at the time of progression.

OUTLINE:

Patients receive lutetium Lu 177 dotatate intravenously (IV) over 30 minutes. Cycles repeat every 6 weeks (Q6W) for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive gallium Ga 68-dotatate IV during screening then undergo positron emission tomography (PET)/computed tomography (CT) scan at baseline and collection of blood throughout the trial.

Patients are followed up at 6 weeks after last dose lutetium Lu 177 dotatate and then every 3 months for 2 years after removal from study or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY
* Patients must have metastatic prostate cancer with neuroendocrine differentiation, as determined by at least one of the following:

  * Histologically confirmed small cell or neuroendocrine cancer from a primary prostate or metastatic biopsy. Neuroendocrine prostate cancer includes mixed small cell with adenocarcinoma histology, as well as small or large cells with positive neuroendocrine markers (e.g., chromogranin or synaptophysin)
  * Prostate adenocarcinoma with molecular features of neuroendocrine differentiated cancer (e.g., 2 of the following 3: PTEN, TP53, or RB loss)
  * Progression of visceral metastases in the absence of PSA progression
  * Serum chromogranin A > 5x normal limit, or neuron-specific enolase > 2x normal NOTE: Both patients who have had prior cytotoxic chemotherapy and patients who have never had cytotoxic chemotherapy for prostate cancer will be allowed
* Age >= 18 years. Prostate cancer is typically a disease of older men, with the average age at diagnosis being 65 years. Consequently, because the research topic is not relevant to children, no children will be included in this study. There is no upper limit to the age of participants eligible for this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8 g/dL, prior to each dose of lutetium lu 177 dotatate
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine Cockcroft calculated creatinine clearance of >= 40 mL/min
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients should be New York Heart Association Functional Classification of class 2B or better
* Current disease progression according to PCWG3 criteria
* Ongoing use of luteinizing hormone-releasing hormone (LHRH) agonists/antagonists will be required (unless prior bilateral orchiectomy or pure neuroendocrine carcinoma histology) to maintain testosterone at castrate levels. Patients with a pure neuroendocrine carcinoma histology do not need to be undergoing LHRH agonist/antagonist therapy
* No concurrent use of other anti-cancer therapies
* Pregnancy Precaution: The effects of lutetium lu 177 dotatate on the developing human fetus are unknown. For this reason and because radionuclides are known to be teratogenic, male participants and their female partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her male partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of lutetium lu 177 dotatate administration. Patients must not donate sperm during the study and for 3 months after the last study drug administration
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Patients will undergo a Gallium 68 Dotatate PET scan after enrollment. The Gallium 68 Dotatate PET must be positive to proceed with lutetium Lu 177 dotatate therapy. A positive scan will be defined as at least one lesion with an maximum standardized uptake value (SUVmax) > the average standardized uptake value (SUV) of normal liver. The positive lesion(s) can be in any location (bone metastases or visceral metastases). Patients with only bone metastases will be allowed
* REGISTRATION ELIGIBILITY: The gallium 68 dotatate PET is positive. A positive scan will be defined as at least one lesion with an maximum standardized uptake value (SUVmax) > the average SUV of normal liver. The positive lesion(s) can be in any location (bone metastases or visceral metastases). Patients with only bone metastases will be allowed.
* REGISTRATION ELIGIBILITY: Absolute neutrophil count ≥ 1,500/mcL
* REGISTRATION ELIGIBILITY: Platelets ≥ 100,000/mcL
* REGISTRATION ELIGIBILITY: Hemoglobin ≥ 8 g/dL, prior to each dose of lutetium Lu 177 dotatate
* REGISTRATION ELIGIBILITY: Total bilirubin ≤1.5 × institutional upper limit of normal (ULN)
* REGISTRATION ELIGIBILITY: AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
* REGISTRATION ELIGIBILITY: Creatinine Cockcroft calculated creatinine clearance of ≥ 40 mL/min OR

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Lutetium Lu 177 dotatate
* As per the Food and Drug Administration (FDA) package insert for Lutetium Lu 177 dotatate, use of long-acting somatostatin analogs (e.g., long-acting octreotide) is prohibited within 4 weeks prior to initiating Lutetium Lu 177 dotatate and during treatment. Use of short-acting somatostatin analogs is prohibited within 24 hours prior to initiating Lutetium Lu 177 dotatate and during treatment. Long-acting somatostatin analogs or short-acting somatostatin analogs will be allowed if the patient has a history of carcinoid syndrome and requires long-acting or short-acting somatostatin analogs for the control of his functional syndrome
* Patients with uncontrolled intercurrent illness
* Any of the following within 6 months before starting treatment: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft; congestive heart failure New York Heart Association (NYHA) Class III or IV
* Uncontrolled hypertension as indicated by a systolic blood pressure >= 160 mmHg or diastolic blood pressure >= 100 mmHg at screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At 6 months
  The objective response rate according to Prostate Cancer Working Group (PCWG) 3 criteria will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). ORR will be reported along with the corresponding two-sided 95% confidence interval. The confidence interval will be adjusted for the two-stage design structure. This analysis will be based on the intent-to-treat population.

SECONDARY OUTCOMES:
Radiographic progression-free survival (rPFS) | At 6 months
  Will be determined by PCWG3 criteria. Specifically, progression/response will be determined via RECIST 1.1 criteria using diagnostic computed tomography (CT) scans of the chest/abdomen/pelvis to analyze progressive disease (PD), stable disease (SD), complete response (CR), partial response (PR), and toxicity type/grade. Progression and response will also be assessed by fludeoxyglucose positron emission tomography (18F-FDG PET).
Treatment response | At 6 months
  Will be assessed by 18F-FDG PET.
Change in FDG-PET signal | Pre-treatment to after 2 doses of lutetium Lu 177 dotatate, assessed up to 16 weeks
  Will be assessed with Quantitative Total Extensible Imaging (QTxI).

OTHER OUTCOMES:
Gene expression levels of circulating tumor cells | Up to 2 years
  Will be summarized using descriptive statistics. Expression levels of candidate markers will be correlated with radiographic time to progression using univariate Cox proportional hazard regression analysis. The Benjamini-Hochberg false discovery rate method will be utilized to control the false discovery rate when evaluating the markers. Machine learning methods will be used to identify signatures of resistance at the time of progression.
Patient-specific dosimetry of lutetium Lu 177 dotatate | Up to 192 hours after first dose of lutetium Lu 177 dotatate
  Descriptive analyses will be conducted to evaluate the potential to perform patient-specific dosimetry of lutetium Lu 177 dotatate using gamma imaging to predict treatment response and renal toxicity. Imaging outcome parameters will be summarized in terms of means, medians, standard deviations and ranges, stratified by assessment time point (24, 96, and 192 hours post-injection), stratified by response (PD, SD versus CR, PR) and toxicity type/grade.

CONTACTS AND LOCATIONS:
Overall Officials: John M Floberg, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (13):
- United States (13):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Northwestern University, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm